CLINICAL TRIAL: NCT07114458
Title: Delirium Incidence and Cognitive Trajectories in Isolated Older Patients in the Inpatient Setting
Brief Title: Delirium and Cognitive Impairment Development in Hospitalized Older Adults Under Isolation Conditions
Acronym: DELiso
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-101313-BO-ff
Record Dates: First submitted 2025-03-16; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Delirium; Dementia; Cognitive Impairment
Keywords: Delirium; neurocognitive disorder; older adult; isolation precautions
MeSH Terms: conditions — Delirium; Dementia; Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposition: Patients under isolation precautions in hospital
- Control: Matched control, no isolation precautions

SUMMARY:
The goal of this observational study is to examine if older patients who need to be under isolation precautions due to multidrug resistant bacteria or other reasons have an increased risk of suffering from delirium or cognitive decline compared to older patients without isolation precautions.

To compare this, every person under isolation precautions is compared to other persons of the same age, gender, comorbidities, frailty status and hospital department. Delirium is assessed twice daily with a screening tool named 3D-CAM and cognitive performance is tested by the MOCA-Test six weeks after discharge from hospital and compared to baseline values which are assessed directly after study enrollment.

The study duration for each patient participating is from the time of enrollment during hospitalization until 6 weeks after hospital discharge.

DETAILED DESCRIPTION:
Delirium is a common complication in older patients during hospitalization. Its prevention is crucial, as it increases morbidity, mortality, and cognitive impairment. Isolation precautions in hospital may further increase delirium risk due to sensory deprivation and reduced mobility.

This study examines the impact of isolation precautions on delirium and neurocognitive disorders in patients ≥70 years. Delirium screening will occur twice daily, with a six-week post-discharge follow-up.

A prospective cohort study will compare delirium incidence in isolated patients with a matched non-isolated control group (matched for age, gender, Charlson Comorbidity Index, Frailty and hospital department). The 3D Confusion Assessment Method (3D-CAM) will be used for Delirium screening. Follow-up assessments will evaluate cognitive function and quality of life. Data will be collected during hospitalization (Days 1-5) and six weeks post-discharge.

ELIGIBILITY:
Inclusion Criteria: - hospitalized patients

* under isolation precautions for at least 24h
* 70 years and above

Exclusion Criteria: - no informed consent

* intensive care treatment
* life expectancy 14 days or less

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospitalized patients of the University Medical Centre Hamburg (all departments)
Sampling Method: Non-Probability Sample
Enrollment: 404 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Delirium | day 1-5 under isolation precautions
  Delirium screened by 3D-Confusion Assessment Method 2 times daily

SECONDARY OUTCOMES:
Cognitive performance | at enrollment and six weeks after discharge from hospital
  Measures by Montreal Cognitive Assessment (MOCA). Maximum 15, minimum 0 points. Higher points indicate less functional impairment.
Functional state | at enrollment and six weeks after discharge from hospital
  Daily activities and functionality assessed by WHO Disability Assessment Schedule (WHODAS 2.0), a questionnaire with 36-items; answers are on a 5-step-Likert-scale; when values are summed up, higher values indicate a worse functional state
Quality-of-Life (QoL) | at enrollment and 6 weeks after discharge from hospital
  QoL assessed by WHO Quality of Life in older adults (WHO-QOL-OLD) questionnaire
Quality-of-Life (QoL) | at enrollment and 6 weeks after discharge from hospital
  QoL assessed by Visual Analogue Scale from EQ-5D-5L questionnaire (no abbreviation); Maximum 100 points, minimum 0 points; more points indicate a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Olotu, Dr., MD, Principal Investigator — University Medical Centre Hamburg, Department of Anaesthesiology

IPD SHARING:
Plan to Share IPD: No